CLINICAL TRIAL: NCT05103683
Title: A Phase 1, First in Human, Dose-Escalation Study of TORL-1-23 in Participants With Advanced Cancer
Brief Title: First in Human Study of TORL-1-23 in Participants With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TORL Biotherapeutics, LLC (Industry)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TORL123-001
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; Ovarian Cancer; Endometrial Cancer; NSCLC
Keywords: claudin6
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Dose Finding - Part 1 (Experimental): TORL-1-23
  Interventions: Drug: TORL-1-23
- Expansion as Monotherapy - Part 2 (Experimental): TORL-1-23
  Interventions: Drug: TORL-1-23

INTERVENTIONS:
Drug: TORL-1-23 — antibody drug conjugate (ADC)

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of TORL-1-23 in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Measurable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Has not recovered [recovery is defined as NCI CTCAE, version 5.0, grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of TORL-1-23
* Progressive or symptomatic brain metastases
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection
* History of significant cardiac disease
* History of myelodysplastic syndrome (MDS) or AML
* History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. A history of other malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ (DCIS) of the breast and prostate cancer with a Gleason score less than or equal to 6, are also not excluded
* If female, is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum Tolerated Dose (MTD) | 28 Days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Time to Response (TTR) | up to 2 years
  Time from start of treatment to complete response or partial response
1 Year Overall Survival (1YOS) | 1 year
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive.
Maximum Serum Concentration of TORL-1-23 (Cmax) | 21 days
  PK assessment
Minimum Serum Concentration of TORL-1-23 (Cmin) | 21 days
  PK assessment
Maximum Serum Concentration of TORL-1-23 at Steady State (Cmax,ss) | 63 days
  PK assessment
Minimum Serum Concentration of TORL-1-23 at Steady State (Cmin,ss) | 63 days
  PK assessment
Time of Maximum Serum Concentration of TORL-1-23 (Tmax) | 21 days
  PK assessment
Time of Minimum Serum Concentration of TORL-1-23 (Tmin) | 21 days
  PK Assessment
Time of Minimum Serum Concentration of TORL-1-23 at Steady State (Tmin,ss) | 63 days
  PK Assessment
Terminal Half-life (t1/2) of Serum TORL-1-23 | 63 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUClast) for TORL-1-23 | 21 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUCinf) for TORL-1-23 | 63 days
  PK Assessment
Apparent volume of distribution during the terminal phase (Vz) of TORL-1-23 | 63 days
  PK Assessment
Clearance (CL) of TORL-1-23 | 63 days
  PK Assessment
Accumulation ratio (Rac) of TORL-1-23 | 63 days
  PK Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Dokainish, Study Chair — TORL Biotherapeutics, LLC
Locations (14):
- United States (9):
  - Providence Medical Foundation, Fullerton, California
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon Research Institute Texas Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- South Korea (5):
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No